CLINICAL TRIAL: NCT02617095
Title: Comparison of the Efficacy and Safety of T2762 Versus Optive® in the Treatment of Moderate to Severe Dry Eye Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment rate too slow
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2762-PIV-11/13
Record Dates: First submitted 2015-11-26; First posted 2015-11-30 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2762 (Experimental): One drop of T2762 in each eye 3 to 6 times daily
  Interventions: Device: T2762
- Optive (Active Comparator): One drop of Optive in each eye 3 to 6 times daily
  Interventions: Device: Optive

INTERVENTIONS:
Device: T2762 — One drop in each eye 3 to 6 times daily
  Arms: T2762
Device: Optive — One drop in each eye 3 to 6 times daily
  Arms: Optive

SUMMARY:
The purpose of this study is to compare the efficacy and safety of T2762 versus Optive® in the treatment of moderate to severe Dry Eye Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Male or female aged ≥ 18 years old.
* Diagnosis of moderate to severe dry eye syndrome

Exclusion Criteria:

* Pregnancy, lactation.
* Childbearing potential woman who is not using a reliable method of contraception and is not surgically sterilised.
* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Non-compliant patient
* Participation in another clinical study at the same time as the present study.
* Participation to the present study during the exclusion period of another clinical study.
* Already included once in this study.
* Ward of court.
* Patient not covered by government health care scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change of the symptomatology evaluation on a Visual Analogic Scale | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Frank Larkin, Professor, Principal Investigator — Moorfields Eye Hospital -162 city road - London; Friedrich KRUSE, Professor, Principal Investigator — Augenklinik mit Poliklinik - Swabachanlage 6 - 91054 Erlangen
Locations (1):
- Laboratoires Théa, Clermont-Ferrand, France